CLINICAL TRIAL: NCT06777446
Title: Elective Adhesiolysis vs. a Wait-and-see Policy to Prevent Recurrences After Conservative Treatment of Adhesive Small Bowel Obstruction
Acronym: AWARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); KCE Belgian Healthcare Knowledge Centre (Unknown); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL88020.091.24
Record Dates: First submitted 2024-12-30; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: Tissue adhesions; Adhesiolysis; Surgery
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Multicenter open-label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Elective Adhesiolysis (Experimental): Elective adhesiolysis is a surgical procedure in which all adhesions in the abdomen are released. Elective adhesiolysis is preferably performed laparoscopy, but the precise surgical approach is adjusted to the expected location and extent of the adhesions based on factors including: presence of a stoma, abdominal wall defects, as well as the surgical history and locations of previous scarring.
  Interventions: Procedure: Elective Adhesionlysis; Device: Adhesion barrier
- Wait-and-see policy (No Intervention): A Wait-and-see policy is the current standard of care after a non-operatively treated epsiode of ASBO. No specific intervention or follow-up is performed in the control group of wait-and-see policy.

INTERVENTIONS:
Procedure: Elective Adhesionlysis — See descriptions in study arms
  Arms: Elective Adhesiolysis
Device: Adhesion barrier — At the end of adhesiolysis a barrier will be placed. The adhesion barrier to be used in laparoscopic adhesiolysis is Icodextrin 4% (Adepttm).
  Arms: Elective Adhesiolysis

SUMMARY:
Rationale: Adhesive small bowel obstruction (aSBO) is a frequent surgical emergency, associated with 3-8% hospital mortality and a high risk of recurrence (20% at two years of follow-up). ASBO can be treated conservatively or by emergency surgery. In the absence of bowel ischemia or strangulation, conservative treatment is often preferred, to avoid the excess morbidity and mortality from emergency surgery. Recent epidemiological studies, however, demonstrate a considerable higher recurrence risk of aSBO after conservative treatment that is associated with hospital readmissions and lower survival. Elective adhesiolysis following successful conservative treatment might reduce these long-term risks whilst avoiding the high complication rate of emergency surgery.

Objective: The investigators aim to assess the efficacy of elective adhesiolysis following conservative treatment for aSBO as compared to the current state of the art (wait-and-see policy) to prevent long-term recurrence of aSBO. Further the investigators will evaluate quality of life, healthcare and societal costs.

Study design: Multicenter open-label randomized controlled trial, including 380 patients.

Study population: Adult patients who recovered from aSBO by conservative treatment. Patients that are inoperable for medical, anaesthesiological or surgical reasons are excluded. Intervention (if applicable): The intervention of investigation is elective adhesiolysis. Adhesiolysis is an abdominal procedure in which all adhesions are cut, and adhesion prevention applied to reduce the risk of adhesion reformation. The intervention is compared to wait-and-see policy (the current standard treatment)

Main study parameters/endpoints: Primary outcome is recurrence, defined as readmission for obstructive systems with aetiology of adhesions confirmed by CT. The investigators hypothesize a 50% reduction in recurrence in the intervention arm. Secondary outcomes are morbidity from surgery, health-related quality of life (EQ5D), healthcare costs and societal costs (iMCQ and iPCQ)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients in the intervention group are exposed to abdominal surgery, which is associated with a moderate risk of minor complications such as wound infection and haemorrhage, and a small risk of severe complications such as iatrogenic bowel injury. According to our hypothesis, a potential benefit is the reduction in the risk of recurrences. Recurrence of aSBO is associated with a risk of readmissions, reinterventions, and also increased long-term mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and older who have recently recovered from aSBO by small bowel obstruction managed by conservative treatment.
* Patients who have previously been operated (high a prior risk of adhesions) are required to have no signs of other causes of bowel obstruction on imaging studies (CT-scan).
* Patients with no previous operation in history (low a prior risk of adhesions) are required to have typical signs for aSBO on imaging studies (abrupt change of bowel calibre, closed loop, or signs of torsion on vessels in the mesentery on CT-scan).

Exclusion Criteria:

* Patient who are unfit for reoperation for surgical, anesthesiological or medical reasons as determined by multidisciplinary team assessment or pre-operative screening
* Patients with active malignancy, reducing life expectancy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
recurrence of ASBO at 2-years of follow-up | 2 years
  Recurrence is defined as a readmission for symptoms of small bowel obstruction, including lower abdominal pain, bloating and nausea with or without vomiting. In addition imaging by CT-scan should not show indications of other causes of bowel obstruction (such as an incarcerated abdominal wall hernia or tumour), which is over 90% accurate for the diagnosis of ASBO.

SECONDARY OUTCOMES:
Recurrence at 5 year | 5 years
  (identified by record linking[BE] or general practitioner data[NL])
Recurrences needing surgery | 2 years and 5 years
  ASBO recurrence requiring emergency surgery
Morbidity from elective adhesiolysis | 90 days
  Composite of:
  * Serious adverse events and complications, graded by Clavien-Dindo score.
  * Intra-operative events (i.e. bowel injury), graded by ClassIntra®
  * ICU admission
  * Reinterventions within 90 days
Health related quality of life | 2 years
  - Health-related quality of life measured by EQ5D
Gastro-intestinal related quality of life | 2 years
  - Gastro-intestinal related quality of life measured by GIQLI
Healthcare costs | 2 years
  measured by modified iMCQ
Societal costs | 2 years
  measured by modified iMCQ
Cost-effectiveness | 2 years and 5 years
  incremental cost-effectiveness ratio, i.e. cost per QALY

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (5):
  - UZ Antwerpen, Antwerp
  - Hôpital Erasme, Brussels
  - UZ Brussel, Brussles
  - UZ Leuven (National Coordinating Center), Leuven
  - Vitaz Sint-Niklaas, Sint-Niklaas
- Netherlands (9):
  - ZGT Almelo, Almelo
  - OLVG Amsterdam, Amsterdam
  - Maasziekenhuis Pantein Boxmeer, Boxmeer
  - St. Jansdal Harderwijk, Harderwijk
  - MaastrichtUMC+, Maastricht
  - RadboudUMC, Nijmegen
  - Laurentius Ziekenhuis Roermond, Roermond
  - St. Franciscus gasthuis Rotterdam, Rotterdam
  - Vie Curie Venlo, Venlo

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: At the end of the experiment and analyses, all data will be stored for 25 years in accordance with GCP regulations.
Access Criteria: Access to individual data will be made available upon reasonable request for academic purposes

REFERENCES:
- [Background] Krielen P, Kranenburg LPA, Stommel MWJ, Bouvy ND, Tanis PJ, Willemsen JJ, Migchelbrink J, de Ree R, Bormans EMG, van Goor H, Ten Broek RPG; ASBO Snapshot Study Group. Variation in the management of adhesive small bowel obstruction in the Netherlands: a prospective cross-sectional study. Int J Surg. 2023 Aug 1;109(8):2185-2195. doi: 10.1097/JS9.0000000000000471. PMID 37288588
- [Background] van den Beukel BAW, Toneman MK, van Veelen F, van Oud-Alblas MB, van Dongen K, Stommel MWJ, van Goor H, Ten Broek RPG. Elective adhesiolysis for chronic abdominal pain reduces long-term risk of adhesive small bowel obstruction. World J Emerg Surg. 2023 Jan 23;18(1):8. doi: 10.1186/s13017-023-00477-9. PMID 36691000